CLINICAL TRIAL: NCT05950672
Title: The Development and Evaluation of a Novel Cat Assisted Training (CAT) Intervention for Youth With Developmental Disabilities and Their Family Cat
Brief Title: Development and Evaluation CAT and Youth
Acronym: CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Megan MacDonald, professor, Oregon State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HE-2022-29; 1R21HD109853-01 (NIH); 5R21HD109853-02 (NIH)
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-06

CONDITIONS: CAT Intervention Group; Control Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAT Intervention Group (Experimental): The experimental group will take part in the CAT intervention (Table 1) after baseline assessments. All cat-training methods will be positive reinforcement based, using owner-approved food, toys and social reinforcers (e.g. petting).
  Interventions: Behavioral: CAT Intervention Group
- CAT Control Group (No Intervention): Control participants will not participate in the CAT intervention. After the completion of the third assessment (end of proposal-related data collection), control participants will be offered the opportunity to participate in cat training classes.

INTERVENTIONS:
Behavioral: CAT Intervention Group — The experimental group will take part in the CAT intervention after baseline assessments. All cat-training methods will be positive reinforcement based, using owner-approved food, toys and social reinforcers (e.g. petting).
  Arms: CAT Intervention Group

SUMMARY:
This R21 provides a multidisciplinary One Health approach to developing and evaluating a novel Cat Assisted Training (CAT) animal assisted intervention (AAI) for early adolescents with developmental disabilities (DD) and their family cat. Cat social behavior and welfare is heavily influenced by human behavior and training, making it highly likely that cats would also benefit from this program. There remains a critical need for further empirical evaluation of AAI practices, especially those that target the specific needs of youth with disabilities. Further extending the development and evaluation of activity-based AAIs beyond those that include dogs and horses also helps address the critical need to consider and include diverse human participants, creating new equitable opportunities for AAI involvement to those who may have access to cats, but not dogs and horses (due to practical, health, cultural, socio-economic, or other personal reasons).

DETAILED DESCRIPTION:
This R21 provides a multidisciplinary One Health approach to developing and evaluating a novel Cat Assisted Training (CAT) animal assisted intervention (AAI) for early adolescents with developmental disabilities (DD) and their family cat. The novel CAT intervention will be a 6-week cat walking and training program for youth 10 - 12 years old. Participants will learn how to respond appropriately to cat body language, practice fear-free and positive reinforcement-based handling, and training skills, and how to fit a harness and walk their cats on leash. For the human participants, skills and behaviors learned during the intervention are expected to promote and support long-term physical activity, social wellbeing, and lasting feelings of responsibility even after the intervention itself has concluded. We also expect these experiences to improve the relationship between the child participant and household cat, and in turn, reduce cat stress in the child's presence and increase cat sociability and indicators of behavioral wellbeing. Because each child will participate with a cat already living in their household, this program will create a unique active partnership between child and cat that considers the health and wellbeing of both partners. Recent pilot work by PIs Udell & MacDonald has revealed physical and social-emotional improvements in children with and without developmental disabilities following a pet dog-partner based AAI. Dogs also showed increased sociability and attachment towards their child partner after AAI participation. Work by PI Udell & Vitale has demonstrated that many cats are highly social and form strong attachment bonds with humans, that cats can be successfully trained a wide range of behaviors, including leash walking, and that cat training classes result in high participant retention rates. Cat social behavior and welfare is also heavily influenced by human behavior and training, making it highly likely that cats would also benefit from this program. There remains a critical need for further empirical evaluation of AAI practices, especially those that target the specific needs of at-risk populations and youth. Further extending the development and evaluation of activity-based AAIs beyond those that include dogs and horses also helps address the critical need to consider and include diverse human participants, creating new equitable opportunities for AAI involvement to those who may have access to cats, but not dogs and horses (due to practical, health, cultural, socio-economic, or other personal reasons).

ELIGIBILITY:
Inclusion Criteria:

* Child with a developmental disability per parental report.
* Family owns a family cat.

Exclusion Criteria:

* Can not follow instructions.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Rate of secure attachment | One year
  A cat sociability and Secure Base attachment test will be conducted to evaluate the cat-child bond (and the cat-adult bond at baseline).

SECONDARY OUTCOMES:
Rate of Physical Activity | One year
  Survey items about pet walking, training and joint activity found on the validated Pet Care Responsibility Inventory will be used to determine if intervention participation predicts a subsequent increase in joint physical activity (including walking and training behaviors) in CAT participants after the intervention,

OTHER OUTCOMES:
Level of Social well being | One year
  Human participants will complete a 1-page Emotional Support survey validated for children ages 8-17.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research will involve a small sample (target N = 30 participants) of youth with DD within a narrow age range recruited from Corvallis and the surrounding counties/ communities. Participants must also have a pet cat to participate in this study. Even with the removal of all identifiers, we believe that it would be difficult to protect the identities of subjects given the small region of recruitment and possible identifying characteristics of subjects and their family cats. Given that some participants may exhibit anxiety, depression or other behavioral and emotional disorders we plan to take every measure to ensure their identify is protected. Therefore, we are not planning to share non-aggregate data.